CLINICAL TRIAL: NCT03046979
Title: Study of Apatinib in Advanced Hepatocellular Carcinoma(HCC)
Acronym: HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBH002
Record Dates: First submitted 2017-01-16; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: apatinib; advanced hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib (Experimental): a molecular targeted anti-tumor drugs. Small molecule vascular endothelial growth factor receptor 2 inhibitor.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500mg, once a day, oral of each 28 day cycle. Number of cycle: until progression or unacceptable toxicity develops.
  Other Names: apatinib mesylate tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of apatinib in patients with advanced HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary malignant tumor of the liver. It is lack of effective drugs for systemic treatment of HCC. Currently, Sorafenib is the only choice approved by FDA for advanced HCC, although it prolongs the survival for less than 3 months. The treatment of advanced HCC still has a long way to go.

At present, the relevant phase II and phase III clinical studies of apatinib on advanced HCC are ongoing. Based on our important discovery of our previous clinical studies, we intends to enlarge the sample size and make further observation for the efficacy and safety of apatinib in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Before doing any research steps, the patient's informed consent must be obtained first.
2. The diagnosis of HCC: histologic diagnosis or Alpha fetoprotein (AFP) with two kinds of imaging diagnosis.
3. Patients of Barcelona stage(BCLC) C with first-line treatment failure or non tolerance to sorafenib.
4. Ages of 18 to 75 years old.
5. Child-Pugh score between 5-7 points, patients of Child-Pugh 7 points should be without ascites.
6. Eastern Cooperative Oncology Group performance score (ECOG PS) is 0-1 point.
7. Adequate organ function meeting the following:

   Hemoglobin(HBG)≧9.0g/dl Neutrophil count(ANC) ≧1,500/mm3 Platelet count(PLT)≧50,000/ul Total bilirubin (TBIL)< 2mg/dL (3mg/dL, Child-Pugh B) Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 5×ULN (upper limit of normal) ALP (alkaline phosphatase ) < 4×ULN PT (prothrombin time) >50% or PT-INR<2.3, <6 seconds or greater than that of the control
8. For patients taking warfarin, at least once a week to a close monitoring of the patients, until, according to the standard of treatment, at every time of medication, the subjects' INR measurements has been stable
9. SCr (serum creatinine) <1.5×ULN
10. For pregnant women, the results of serum pregnancy tests must be negative within 14 days before initiation of treatment.
11. All men and women who participated in the study had to take reliable contraceptive measures within the trial and two weeks of after the trial.

Exclusion Criteria:

1. Patients of Child-Pugh 7 has serious uncontrolled ascites.
2. Patients with serious cardiovascular disease.
3. Patients with high blood pressure of unable to control.
4. Patients has the history of HIV (human immunodeficiency virus) infection.
5. Active clinical severe infection (> 2, NCI-CTCAE version 3).
6. Need to drug treatment of patients with epilepsy (such as steroid or antiepileptic drugs)
7. Has a history of allogeneic organ transplantation.
8. Patients with a history of physical signs or have a bleeding.
9. Patients undergoing renal dialysis.
10. Metastatic liver cancer.
11. Patients with uncontrollable ascites.
12. Patients with encephalopathy.
13. Patients has history of gastrointestinal bleeding period of 30 days before join the study.
14. Patients with a history of esophagus varicosity burst hemorrhage, then not effective treatment or therapy to prevent recurrence of bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | one year

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | one year
Progression free survival (PFS) | one year
Overall survival (OS) | one year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0[Quality of life] | one year
Incidence of Treatment-Emergent Adverse Events [Safety] | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ti Zhang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided
the plan to share IPD is under consideration.

REFERENCES:
- [Derived] Hou Z, Zhu K, Yang X, Chen P, Zhang W, Cui Y, Zhu X, Song T, Li Q, Li H, Zhang T. Apatinib as first-line treatment in patients with advanced hepatocellular carcinoma: a phase II clinical trial. Ann Transl Med. 2020 Sep;8(17):1047. doi: 10.21037/atm-20-2990. PMID 33145266